CLINICAL TRIAL: NCT02325596
Title: Investigate the Role of microRNA in Chronic Rhinosinusitis From DC-Th Axis
Acronym: ITROMICRFDTA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Guo-hua Hu, Investigate the Role of microRNA in Chronic Rhinosinusitis From DC-Th Axis, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: NSFC-81271061
Record Dates: First submitted 2014-12-15; First posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Rhinosinusitis
Keywords: Chronic rhinosinusitis; microRNA; dendritic cell; helper T cell
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- control: Patients with only nasal septum deviation
  Interventions: Genetic: miRNA mimics or inhibitors
- CRS sNP: Chronic Rhinosinusitis patients without nasal polyps
  Interventions: Genetic: miRNA mimics or inhibitors
- atopic CRS wNP: Chronic Rhinosinusitis patients with allergic constitution and nasal polyps
  Interventions: Genetic: miRNA mimics or inhibitors
- non-atopic CRS wNP: Chronic Rhinosinusitis patients with nasal polyps but not allergic constitution
  Interventions: Genetic: miRNA mimics or inhibitors

INTERVENTIONS:
Genetic: miRNA mimics or inhibitors — DCs are transfected by the miRNA mimics or inhibitors after they are separated from peripheral blood mononuclear cells in CRS patients

SUMMARY:
This study aimed to evaluate the upstream events of Th17/Treg imbalance in CRS and their immune regulatory factors. Then the investigators aimed to explore the regulatory role of miRNA on DC-Th axis and its dysfunction in the pathogenesis of CRS, in order to determine the miRNA expression profile in CRS and clarify the role of miRNA in the pathogenesis of CRS by regulating the DC-Th axis.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS), commonly encountered in the ﬁeld of clinical otorhinolaryngology, is still a challenging proposition for doctors because of its high incidence and the unsatisfactory treatment outcomes. Nowadays, studies on the pathogenesis of NP are still attached great importance by researchers from each country. NP has become a global health problem with a considerable socioeconomic burden. Recently, research showed that the impaired balance of Th17/Treg was the significant basis of NP. Nevertheless, the pathogenesis of Th17/Treg imbalance was unclear. In this study, DC-Th axis was designed as the main line, and the regulation of miRNA on DC was designed as the entry point. This study aimed to evaluate the upstream events of Th17/Treg imbalance in CRS and their immune regulatory factors. Then the investigators aimed to explore the regulatory role of miRNA on DC-Th axis and its dysfunction in the pathogenesis of CRS, in order to determine the miRNA expression profile in CRS and clarify the role of miRNA in the pathogenesis of CRS by regulating the DC-Th axis. This study will play an important role in clarifying the pathogenesis of CRS eventually and will fill the blanks of the research between miRNA and CRS in the investigators'country. This study is with important clinical value for establishing control strategies for CRS.

ELIGIBILITY:
Inclusion Criteria:

1. CRS diagnosis is accord with diagnostic criteria of The European nasal sinusitis, nasal polyps guidelines (EPOS 2012) .
2. Selected subjects are stopped using systemic or topical corticosteroids in one month before experiment.
3. All the patients have sinus CT and nasal endoscopy and allergen Skin Prick Test in preoperative.
4. Aged from 18 to 75 years old.
5. Woman or man.

Exclusion Criteria:

1. Choanal polyp, fungal nasal sinusitis, cystic fibrosis.
2. Acute upper respiratory tract infection and other diseases associated with the body.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the department of endoscopic sinus surgery in the First Affiliated Hospital of Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Abnormal microRNA in the Chronic Rhinosinusitis are found by gene chip and qPCR. | 6 to 24 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guo-hua Hu HG Guo-hua Hu, MD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Ma ZX, Tan X, Shen Y, Ke X, Yang YC, He XB, Wang ZH, Dai YB, Hong SL, Hu GH. MicroRNA expression profile of mature dendritic cell in chronic rhinosinusitis. Inflamm Res. 2015 Nov;64(11):885-93. doi: 10.1007/s00011-015-0870-5. Epub 2015 Sep 4. PMID 26337346